CLINICAL TRIAL: NCT05983146
Title: A Phase I, Open-label, Multi-center Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of HRS-7053 Injection in Patients With Advanced Malignancies
Brief Title: Phase I Study of HRS-7053 Injection in the Treatment of Patients With Advanced Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor's R&D strategy is adjusted.
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7053-101
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignant Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-7053 Injection (Experimental)
  Interventions: Drug: HRS-7053 Injection

INTERVENTIONS:
Drug: HRS-7053 Injection — HRS-7053 is administered by intravenous (IV) infusion once a week (QW) for one treatment cycle every 4 weeks

SUMMARY:
To evaluate the safety and tolerability of multiple administration of HRS-7053 in patients with advanced malignancies Determine the maximum tolerated dose (MTD, if possible) and the recommended dose for Phase II clinical studies (RP2D)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this study, signed informed consent, compliance is good, can cooperate with follow-up
2. Age ≥18 years, both male and female
3. Histologically or cytologically confirmed patients with advanced hematologic malignancies that have not responded to standard antitumor therapy and currently indicate treatment
4. Have measurable lesions
5. ECOG PS score: 0-1
6. Have a life expectancy of at least 3 months
7. The functional level of the major organs must meet the requirements
8. Fertile female patients must have a serum pregnancy test within 7 days before the first medication and the result is negative; And must be non-lactating

Exclusion Criteria:

1. The tumor infiltrates the central nervous system
2. Received autologous stem cell transplantation within 12 weeks prior to administration of the first study; Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation; In the first study, Car T cell therapy was administered within 12 weeks prior to drug administration
3. Had major surgery or severe trauma 4 weeks prior to the first study; Or plan to undergo major surgery during the study
4. Received antitumor therapy within 2 weeks prior to administration of the first study drug; Received Chinese herbal therapy within 2 weeks before the first dose of study drug administration; Receiving steroid hormones for antitumor purposes within 7 days before the first dose of the investigational drug administration
5. Use of live attenuated vaccine within 28 days prior to signing the informed consent, or expected to require live attenuated vaccine during the study period to 5 months after the final dose
6. Use of any potent drug that inhibits the liver drug metabolizing enzyme CYP3A for 14 days prior to first administration; Any potent drug that induces the liver drug metabolizing enzyme CYP3A has been used for 28 days prior to first administration
7. Previous treatment-induced adverse events did not recover to ≤CTCAE grade 1
8. Participating in other clinical studies or signing informed consent less than 1 month after the last medication in the previous clinical study
9. The active phase of HBV or HCV infection is known
10. A history of immunodeficiency, including HIV seropositive, or other acquired, congenital immunodeficiency disorders
11. Active infection or unexplained fever > 38.5 ° c
12. A history of clinically severe cardiovascular disease; A history of myocarditis within one year prior to drug administration was first studied
13. The abnormality of electrocardiogram (ECG) was clinically significant
14. In the first study, cerebrovascular accident, transient ischemic attack occurred within 6 months prior to drug administration
15. History of other malignancies within 5 years prior to drug administration was first studied
16. Known allergy to any component of the HRS-7053 product
17. The presence of other serious physical or mental illnesses, abnormal laboratory tests, and other factors that may increase the risk of participating in the study or interfere with the study results; And any other conditions that the investigator deems inappropriate for participation in this study
18. Female subjects are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AES) | up to 3 years
MTD | up to 3 years
RP2D | up to 3 years

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | up to 3 years
Maximum concentration (Cmax) | up to 3 years
Area under the time curve from 0 to the last measurable concentration time point t (AUC0-t) | up to 3 years
Objective response rate （ORR） | up to 3 years]
Disease control rate (DCR) | up to 3 years
Progression-free survival (PFS) | up to 3 years
Duration of response (DoR) | up to 3 years
Overall survival (OS) | up to 3 years

IPD SHARING:
Plan to Share IPD: Undecided